CLINICAL TRIAL: NCT02604238
Title: Efficacy and Safety of Thrombolytic Therapy With Half Dose Alteplase, Added to Standard Anticoagulation Therapy With Heparine, in Patients With Moderate Pulmonary Embolism: a Prospective, Randomized, Open Label,Controlled Trial
Brief Title: Efficacy and Safety of Half Dose Alteplase Added to Heparine, in Patients With Moderate Pulmonary Embolism
Acronym: MONALYSE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda U.S.L. 1 di Massa e Carrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Azienda USL1 Massa e Carrara
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism at intermediate risk
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Administered a "safe dose" of Alteplase. All patients are treated with low molecular weight heparin ( LMWH ) according to the Guidelines ESC2014 heparin in addition it is administered a "safe dose" of Alteplase.
  Interventions: Drug: Alteplase
- Group B (No Intervention): All patients are treated with low molecular weight heparin ( LMWH ) according to the Guidelines ESC2014 heparin. It not added any treatment.

INTERVENTIONS:
Drug: Alteplase — Enoxaparin (1mg) 100UI aXa/kg/sc [LMWH], 15 -30 minutes prior to administration of intravenous (iv) bolus loading dose of 10 mg in 1 min, followed by iv infusion of 40 mg within two hours (for patients weighing <50 kg, a loading dose of bolus of 0.5 mg in 1 min, followed by iv infusion of 40 mg in two hours); the infusion will be adjusted to maintain the value of aPTT between 50-70 seconds (1.5 to 2.5 times the reference value).
  Other Names: tPA-tissue Plasminigen Activator
  Arms: Group A

SUMMARY:
The primary aim of this study is to evaluate whether mid dose (safe dose) of Alteplase in addition to standard treatment with heparin (LMWH) in patients with pulmonary embolism (PE) at intermediate risk, it is effective to reduce:

* right ventricular dysfunction
* pulmonary hypertension 24 hours and 7 days after the treatment
* PE recurrence to 7days and 30 days after the treatment without increasing the incidence of bleeding intra-extracranial

DETAILED DESCRIPTION:
The guidelines of the European Society of Cardiology (ESC2014) confirm the indication for pharmacological revascularization with thrombolysis only to cases of pulmonary embolism at high risk and thus hemodynamically unstable (class of recommendation I, level of evidence B), reserving the surgical or interventional procedures to cases where thrombolysis has failed or is contraindicated, while it remains controversial the role of thrombolysis in patients with pulmonary embolism at intermediate risk; the current state, in EP intermediate risk, the standard treatment involves the administration of low molecular weight heparin (LMWH), or fondaparinux (for 5-10 days followed by anticoagulation therapy with vitamin K antagonists) or alternatively the new anticoagulants oral (NAO). Although the results of the study PEITHO, recently published, confirm the indication for thrombolytic therapy for primary reperfusion in patients with embolism pulmonary high risk and provide element of reflection about the incidence of intracranial hemorrhage major, recent studies suggest that the thrombolysis with tPA to reduced dose (about half the dose that used in standard thrombolysis) in addition to anticoagulants (low molecular weight heparin) may reduce pulmonary hypertension (systolic artery pulmonary pressure> 40 mmHg) and the incidence of recurrent PE. In this protocol, based on the study MOPETT and pharmacokinetic data available, it is used a "safe dose" (safe dose reduced) of alteplase which provides a intravenous (iv) bolus loading dose of 10 mg in 1 min, followed by intravenous infusion 40 mg within two hours (for patients weighing <50 kg loading dose iv bolus of 0.5 mg in 1 min, followed by iv infusion of 40 mg within two hours).

After treatment with alteplase, the heparin therapy will be resumed when aPTT values are less than twice the upper limit of normal; the infusion will be adjusted to maintain aPTT between 50-70 seconds (1.5 to 2.5 times the reference value), and for safety reasons are excluded patients> 65 -70 years (increased risk of bleeding complications related age and comorbidities).

ELIGIBILITY:
Inclusion Criteria:

1. pulmonary embolism at intermediate risk as defined by the Guidelines ESC2014[ documented pulmonary CT angiography]
2. pulmonary hypertension (systolic pulmonary pressure greater or equal to 40 mm Hg) [documented echocardiogram presence of thrombotic material in the right-sided]
3. disfunction Ventricular right confirmed by echocardiogram or TC chest:

   * dilation of the right sections (> 30 mm in parasternal or relationship right ventricle/left ventricle > 1)
   * paradoxical movement of the interventricular septum
   * TAPSE reduced (Tricuspid Annular Plane Systolic Excursion)
   * tricuspid regurgitation with gradient VD/AD> 30 mmHg, in the absence of right ventricular hypertrophy, McConnell sign (apical segment of the free wall of the right ventricle normalKinetic or hyperkinetic than a hypokinesia or akinesia of the remaining parts of the right ventricular wall),
4. myocardial damage confirmed with:

   * Troponin I or T positive
   * higt value of the biomarkers of myocardial damage : BNP or NTproBNP
5. informed consent

Exclusion Criteria:

1. age <18 years and> 65 years
2. HASBLED score ≥ 3 (23)
3. intracranial tumors
4. ischemic stroke within 2 months
5. surgery neurological within 1 month and surgery within 10 days
6. trauma within 15 days
7. hypotension to hospitalization (systemic blood pressure <90 mmHg)
8. uncontrolled hypertension (SBP> 180mmHg and PAD> 110mmHg)
9. clotting disorders
10. thrombocytopenia (<100.000)
11. platelet counts below 100 × 109 /L severe thrombocytopenia (platelet count <50.000 ptl / mm3)
12. liver failure
13. kidney failure
14. gastrointestinal bleeding within 10 days
15. pregnancy or childbirth within 30 days
16. contraindications to the use of thrombolytics
17. contraindications to the use of low molecular weight heparin (enoxaparin)
18. anticoagulation therapy started more than 8 hours
19. COPD
20. endocarditis
21. severe obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary hypertension reduction (systolic pulmonary pressure greater or equal to 30 mm Hg) | 24 hour
  Pulmonary hypertension reduction documented on echocardiography

SECONDARY OUTCOMES:
Incidence of recurrent pulmonary embolism fatal or non fatal | 7 days
  Incidence of recurrent pulmonary embolism fatal or non fatal
Incidence of hemodynamic shock | 24 hour and 30 days
  Incidence of hemodynamic shock [defined as: need for cardiopulmonary resuscitation, or SBP <90 mmHg for a period ≥15 min or reduction SBP ≥40 mm Hg for SBP ≥15 min, with evidence of systemic hypoperfusion (cold extremities, diuresis <30 mL / h, mental confusion), or need for infusion of amines to maintain adequate organ perfusion and SBP> 90 mm Hg
Incidence of hospital death from all causes | 30days
  Incidence of hospital death from all causes

OTHER OUTCOMES:
Bleeding extracranial minor and major | 24 hour and 30 days
  Bleeding extracranial minor and major

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Conti, MD, Principal Investigator — Azienda USL1 di Massa e Carrara